CLINICAL TRIAL: NCT06663501
Title: Effects of Vibration on Motor Function of Survivors of Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Zev Rymer, Director Single Motor Unit Laboratory, Shirley Ryan AbilityLab
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00219884
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Healthy
Keywords: Upper extremity; AMES; Proprioception; Vibration
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single-site exploratory, unrandomized, the first arm is persons with stroke, the second arm is uninjured controls. Both Cohorts receive the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stroke Intervention (Experimental): In this arm, the participant will be scheduled to come to the laboratory 2-4 times per week and spend 30 minutes using the Assisted Motion with Enhanced Sensation (AMES) treatment device on the affected side of the upper limb.
  Interventions: Device: Assisted Motion with Enhanced Sensation training
- Uninjured Control Intervention (Active Comparator): In this arm the uninjured controls will perform the same interventions as the stroke group. The uninjured control group will perform the tests and interventions with their dominant arm/hand.
  Interventions: Device: Assisted Motion with Enhanced Sensation training

INTERVENTIONS:
Device: Assisted Motion with Enhanced Sensation training — During the AMES intervention, the AMES device will flex or extend the wrist/hand joint, and the participant's task will be to assist this motion. As the wrist/hand joint moves, the machine will be delivering a vibratory mechanical stimulus on the opposite side to the direction of movement. The activity of the muscles during the movement of the wrist/hand joint will be recorded by the device and it will be shown on a screen to be used as feedback during the training
  Other Names: AMES Training

SUMMARY:
The aim of this study is to evaluate how vibration of the tendons enhances arm and hand training in survivors of chronic stroke.

The investigators hypothesize that wrist/elbow robotic training, combined with body awareness training will improve arm and hand function in individuals with chronic stroke.

DETAILED DESCRIPTION:
Each year, more than 600,000 U.S. citizens experience a major stroke. Following acute care, 30-40% of these survivors sustain permanent motor disabilities. The motor symptoms of stroke include loss of muscle control on one side of the body, spasticity, and loss of coordination ("dyssynergia"). Within days of the stroke, surviving patients begin physical therapy to restore motion, with some recovering completely. However, there are over 5 million individuals in the U.S. alone who have not recovered and are severely incapacitated for the remainder of their lives. Recovery of function typically reaches a plateau within 6-12 months following a stroke. This recovery of function presumably involves "plastic" changes in the cerebral cortex, in which new neural circuits organize to replace those damaged by the injury. The origin of paralysis or paresis (i.e., partial loss of movement) and the cause of spasticity are unclear in many stroke patients. In a small subset, the brain tissue injured by the stroke is localized to the "primary motor cortex", which contains the nerve cells that send movement signals to the muscles. Loss of movement is easy to understand in these individuals. However, in many strokes, the injury is located in other parts of the brain or is more diffuse, and loss of movement is not as easy to explain. In many regions of the brain, sensory information from various sources, including the proprioceptive system, is integrated and then relayed to the motor cortex to produce movement.

Proprioception is the sense of body position and movement, which originates from sensory receptors in muscles, tendons, skin, and joints. Research carried out over the last two decades indicates that proprioception is intimately involved in motor coordination. In fact, individuals who suffer a rapid loss of proprioception they are functionally paralyzed for a period of time. The hypothesis underlying our approach to stroke rehabilitation is that, in many survivors of stroke, the damage to the brain disrupts one or more feedback loops that connect the proprioceptive receiving areas of the primary somatosensory cortex (Areas 1, 2, 3a, and 3b) to the primary and pre-motor cortex (Areas 4 and 6). Without proprioceptive information feeding into the motor output center, the brain cannot "locate" the muscles needed for movement to occur. We hypothesize that the synchronous and repetitive activity of the input and output areas of the cortex stimulates the reorganization of the brain pathways, thereby closing the feedback loop(s) disrupted by the stroke. In this context, the aim of our research is to identify the effect of a wrist/elbow robotic assisted training combined with proprioceptive training provided by repetitive vibratory stimuli in the tendons of the muscles involved in wrist/elbow flexion and extension on voluntary movement like the reaching movements in individuals with chronic stroke.

In this approach to stroke rehabilitation, the investigators aim to enhance plastic changes in the brain following the injury by repetitively causing the nerve cells in the primary somatosensory cortex to fire synchronously with nerve cells in the functionally related parts of the motor cortex. This approach is designed to rebuild the connections between incoming proprioceptive input and outgoing motor output.

The research objective is to develop procedures to rehabilitate participants > 1 year post-stroke who, through conventional therapies, are not brought to a level of maximal recovery. The aim of the proposed project is to obtain a set of data from a total of 20 chronic stroke participants, all with severe upper extremity disability, between the ages of 18-85, using a robotic therapeutic device placed in a biomechanics laboratory within the Shirley Ryan AbilityLab. This data will allow us to quantify the extent to which a combination of robotic-assisted exercise and tendon vibration induces secondary recovery from stroke in the upper extremity.

The proposed research plan involves a machine with 2 main components, a range of motion sensor and sensory stimulators (i.e., mechanical vibrators). The range-of-motion component of the machine rotates the affected joint (e.g., wrist or elbow) and records position and force. The participant's task involves contracting muscles to assist with the applied motion. Visual feedback of the amount of force or Electromyographic (EMG) activity produced by the participant is displayed on a computer screen. The assisted movement activates the nerve cells in the motor cortex of the brain. While the combined efforts of the robotic device and the participant repeatedly rotate the participant's paretic wrist/elbow into flexion and extension, a pair of vibrators delivers high frequency stimulation (60 pulses per second) to the corresponding tendons on the side of the joint opposite to the agonist muscles. Vibration is known to be an effective stimulus for muscle spindles, the primary sensory receptors that contribute to proprioception. The vibration stimulus increases, by several-fold, the natural response of the muscle spindles to the joint rotation. Only the lengthening tendon is vibrated at any given time. The vibration-induced activation of muscle spindles in the lengthening muscle(s) serve to activate the nerve cells in the somatosensory cortex of the brain. Thus, assisted exercise activates nerve cells in the motor output area of the cortex while vibration simultaneously activates the functionally related nerve cells in the sensory input area, providing a stimulus to develop new, or to enhance existing connections between the two areas.

ELIGIBILITY:
Inclusion Criteria:

* If stroke, more than 6 months after
* Medically stable
* Not currently taking any anti-spasticity medications (for at least 2 weeks)
* Able to comply with study requirements

Exclusion Criteria:

* Recent change in the use of any medications
* Other physical conditions such as orthopedic injuries or surgeries
* Unstable Medical conditions or any other clinical observations that may affect the candidates performance, health, safety, or ability to participate in the study as determined by the treating therapist
* Anti-spasticity drug injection in the 3 months prior to participation
* Presence of significant cardiorespiratory or metabolic disease
* Inability to achieve standard position required for EMG recordings
* Intrathecal baclofen pump
* Musculoskeletal conditions/surgeries resulting in difficulty participating
* Adults unable to consent
* Pregnant women, prisoners, and individuals under the age of 18

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment for the upper extremity score | 1 day following intervention
  The Fugl-Meyer Assessment for the upper extremity measures the severity of injury following a stroke. The assessment is scored from 0-66 points. A higher score indicates less impairment

SECONDARY OUTCOMES:
Proprioception Assessment | 1 day following intervention
  Using the AMES device, proprioception (wrist/elbow position sensing), is assessed, while blindfolded, the participant will be moved to a specific angular position then back to neutral. The participant will be asked to voluntarily move the joint back to the earlier position without vision
Modified Ashworth Score | 1 day following intervention
  An assessment of spasticity of the upper extremity. This is scored from 0-4, with 4 indicating an immobilized joint
Strength Assessment | 1 day following intervention
  Using the AMES device, a load cell will measure the maximum force produced by the wrist or elbow

CONTACTS AND LOCATIONS:
Overall Officials: William Z Rymer, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No